CLINICAL TRIAL: NCT04300348
Title: Real-time Auditory Feedback for Improving Gait and Walking in People With Parkinson's Disease
Brief Title: Improving Walking With Heel-To-Toe Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-5842
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Parkinson
Keywords: gait; walking capacity; neuroplasticity; motor learning; quality of life

STUDY DESIGN:
Intervention Model Description: Standard two-group, sequential design, with 2:1 randomization (intervention:control) and only a within-group analysis.
Who Masked: Outcomes Assessor
Masking Description: An evaluator who does not know to which group the participant was assigned will conduct the evaluations. The outcomes are tests of performance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heel2Toe Group (Active Comparator): The Heel2Toe group will have 5 therapy sessions to learn to trigger the sensor with a strong heel strike and how to use device for home practice for 3 months. During the home practice, participants will be instructed to walk with the device for a minimum of 10 minutes per day in feedback mode. They will be provided with a workbook outlining simple exercises targeting functions needed to walk well (Walk-BEST Workbook) in paper and as a mobile app.
  Interventions: Device: Heel2Toe
- No-feedback Control Group (Control group) (Other): The Control group will do the same 5 sessions of training and 3 months of practice but without the Heel2Toe device in feedback mode, just in data acquisition mode. They will be provided with a workbook outlining simple exercises targeting functions needed to walk well (Walk-BEST Workbook) in paper and as a mobile app.
  Interventions: Other: No-feedback control group

INTERVENTIONS:
Device: Heel2Toe — Heel to Toe (Heel2Toe) is a device that clips on the shoe and provides an instant auditory feedback (a beep) for each correct step characterized by putting the heel first and it provides data on gait parameters
  Arms: Heel2Toe Group
Other: No-feedback control group — The control group will follow the same protocol as the Heel2Toe group but the device will not be in feedback mode just in data acquisition mode.
  Arms: No-feedback Control Group (Control group)

SUMMARY:
Introduction: The purpose of this study is to test the efficacy potential of using real-time positive auditory feedback to improve gait pattern in people with Parkinson's Disease (PD). The components of walking are commonly affected in patients with PD. Gait training for PD is usually based on verbal cues from the therapist that are only moderately effective. Based on good principals of gait and neuroplasticity, the Heel-To-Toe (Heel2Toe) sensor was developed to provide real-time auditory feedback during walking training. Methods: A two-group, randomized feasibility trial is planned with repeated measures of gait parameters and walking outcomes. Participants will be assessed at baseline, 3 and 6 months. Outcomes after the 5 training days will be obtained directly from the Hee2Toe device for both groups (with and without auditory feedback). The primary outcome is walking capacity measured by the Six-Minute Walk Test and the Standardized Walking Obstacle Course. Gait parameters will be captured by the Heel2Toe device Expected Contributions: Gait training using the Heel2Toe sensor will be potentially effective for improving walking pattern in people with PD.

DETAILED DESCRIPTION:
As this is a feasibility study, the main analysis will focus on within-group change over the intervention period of 3 months using indices of reliable change(36). This method assesses the number of people who changed in each of the groups based on the magnitude of change relative to pre-post variability and correlation. We will estimate the proportion of people with reliable change. Estimates from the pilot study will be used to plan the main trial if the pilot demonstrates feasibility. For the maintenance period, reliable change from baseline will also be estimated and used to identify the proportion of people who maintained reliable change or who gained/lost this status.

The study is designed to detect a minimal important within-group change of moderate magnitude or greater (effect size ½ standard deviation) with adequate precision. A sample size of 20 in the intervention with completed follow-up will provide a 95% confidence interval with precision that excludes an effect size of 0.03.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson Disease and be independent in ambulation without use of walking aid

Exclusion Criteria:

* exercising three or more time per week;
* Had any additional illness that restricted their function
* Showing difficulty reading, understanding or speaking either French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Reliable Change in Six-Minute Walk Test | Baseline, 3 months (Change from Baseline to 3 months; maintenance to 6 months)
  Performance-rated outcome
Change in Standardized Walking Obstacle Course (SWOC) | Baseline, 3 months (Change from Baseline to 3 months; maintenance to 6 months)
  Performance-rated outcome of challenges experienced with starting, stopping, turning, making motor decisions. The metric is the time to complete a 12.2-m long, 0.92-m wide curved pathway, with obstacles commonly encountered in daily life.

SECONDARY OUTCOMES:
Safety (Falls) | Baseline to 3 months.
  Self-reported number of falls during study period
Technology acceptability (System Usability Scale) | 3 months (1 time point)
  Patient-reported outcome on satisfaction and intent-to-use
Change in Gait Quality (Data capture from Heel2Toe sensor) | Baseline, 3 months (Change from Baseline to 3 months; maintenance to 6 months)]
  Technologically-reported outcome
Change in Lower Extremity Function (Neuroqol) | Baseline, 3 months (Change from Baseline to 3 months; maintenance to 6 months)
  Patient-reported outcome on degree of difficulty with activities related lower extremity function
Change in Postural Instability and Gait Dysfunction (UPDRS) | Baseline, 3 months (Change from Baseline to 3 months; maintenance to 6 months)
  Self-reported outcome of limitations
Change in health-related quality of life (EQ-5D-3L) | Baseline, 3 months (Change from Baseline to 3 months; maintenance to 6 months)
  Patient-reported outcome (EQ-5D-3L)
Change in motivation (Starkstein Apathy Scale, Activity Effort Inventory) | Baseline, 3 months (Change from Baseline to 3 months; maintenance to 6 months)
  Patient-reported outcome
Change in health states (Visual Analogue Health States) | Baseline, 3 months (Change from Baseline to 3 months; maintenance to 6 months)
  Patient reported outcome of 8 health states measured on 0 to 10 scale
Cognitive performance (Symbol Digit Modality Test) | Baseline, 3 months, 6 months
  Performance-rated outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Mayo, PhD, Principal Investigator — Research Institute - MUHC
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mate KKV, Abou-Sharkh A, Morais JA, Mayo NE. Putting the best foot forward: Relationships between indicators of step quality and cadence in three gait vulnerable populations. NeuroRehabilitation. 2019;44(2):295-301. doi: 10.3233/NRE-182595. PMID 30856128
- [Background] Mate KK, Abou-Sharkh A, Morais JA, Mayo NE. Real-Time Auditory Feedback-Induced Adaptation to Walking Among Seniors Using the Heel2Toe Sensor: Proof-of-Concept Study. JMIR Rehabil Assist Technol. 2019 Dec 11;6(2):e13889. doi: 10.2196/13889. PMID 31825320
- [Background] Carvalho LP, Mate KKV, Cinar E, Abou-Sharkh A, Lafontaine AL, Mayo NE. A new approach toward gait training in patients with Parkinson's Disease. Gait Posture. 2020 Sep;81:14-20. doi: 10.1016/j.gaitpost.2020.06.031. Epub 2020 Jun 29. PMID 32650238
- See also: Website for the company that produces Heel2Toe(TM) — http://physiobiometrics.com